CLINICAL TRIAL: NCT02791009
Title: Asian neTwork for Translational Research and Cardiovascular Trials ("ATTRaCT")
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other); National University Hospital, Singapore (Other); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2194
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: HF; HFrEF; HFpEF; MRI; biomarker
MeSH Terms: conditions — Heart Failure | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specific biomarker profiles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Diagnosed Heart Failure [Prior]: Patients will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI), Cardiovascular Ultrasound (CVUS), Electrocardiogram (ECG), Blood Sample Collection and Clinical Assessment.
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (CMRI); Other: Electrocardiogram (ECG); Other: Blood Sample Collection; Other: Clinical Assessment; Other: Cardiovascular Ultrasound (CVUS)
- Control [Prior]: Control will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI), Cardiovascular Ultrasound (CVUS), Electrocardiogram (ECG), Blood Sample Collection and Clinical Assessment.
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (CMRI); Other: Electrocardiogram (ECG); Other: Blood Sample Collection; Other: Clinical Assessment; Other: Cardiovascular Ultrasound (CVUS)
- Control [New]: Control will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI), Cardiovascular Ultrasound (CVUS), Electrocardiogram (ECG), Blood Sample Collection and Clinical Assessment.
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (CMRI); Other: Electrocardiogram (ECG); Other: Blood Sample Collection; Other: Clinical Assessment; Other: Cardiovascular Ultrasound (CVUS)
- Diagnosed Heart Failure [New]: Patients will undergo the following studying procedures: Cardiovascular Magnetic Resonance Imaging (CMRI), Cardiovascular Ultrasound (CVUS), Electrocardiogram (ECG), Blood Sample Collection, Cognitive Test and Clinical Assessment.
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging (CMRI); Other: Electrocardiogram (ECG); Other: Blood Sample Collection; Other: Clinical Assessment; Other: Cardiovascular Ultrasound (CVUS); Other: Cognitive Test

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imaging (CMRI) — CMRI uses interaction of the magnetic properties of body tissues with strong magnetic fields to create images; for about 1 hour. Several sets of images are needed. No injection of drug or dye will be used for this procedure.
Other: Electrocardiogram (ECG) — ECG is a non-invasive test used to detect any underlying heart conditions by measuring the electrical activity of the heart.
Other: Blood Sample Collection — Blood will be drawn for circulating biomarkers, which are measurable indicators of the severity or presence of the heart failure condition.
Other: Clinical Assessment — Check health status, blood pressure, heart rate, height and weight measured. In addition, subject will undergo a heart examination.
Other: Cardiovascular Ultrasound (CVUS) — To measure heart chamber size, heart function, blood vessel size and blood vessel function. These measurements will help the investigators understand the type and severity of heart failure.
Other: Cognitive Test — To relate the presence and severity of cognitive impairment (CI) with simultaneously acquired advanced cardiovascular imaging characteristics and circulating biomarkers of cardiovascular function, inflammation and coagulation.
  Groups: Diagnosed Heart Failure [New]

SUMMARY:
To build on Singapore's competitive advantages in advanced cardiac imaging, genetic and molecular studies to develop an integrated "one -stop" platform spanning from human to large and small animal models, dedicated to deepening the understanding of CV disease progression, discovery of new targets and repurposing of drugs.

DETAILED DESCRIPTION:
Heart failure (HF) is the final common pathway of cardiovascular (CV) diseases and leading cause of CV hospitalizations in Singapore and worldwide, with a mortality rate that rivals most cancers (>50% mortality at 5 years). Also similar to cancer, HF is a staged disease where early detection and treatment are vital for prevention of disease progression from Stage A (risk factors) to Stage B (subclinical structural heart disease) and Stage C (symptomatic HF). Cardiac imaging is critical for the detection of early subclinical disease. There is limited understanding of the mechanisms underlying disease progression and effective therapies are limited, particularly for the half of the HF population with preserved ejection fraction (HFPEF or "diastolic HF") for which there is no effective therapy to date (in contrast to HF with reduced ejection fraction [HFREF] or "systolic HF").

The investigators overall aim is to build on Singapore's competitive advantages in advanced cardiac imaging, genetic and molecular studies to develop an integrated "one -stop" platform spanning from human to large and small animal models, dedicated to deepening the understanding of CV disease progression, discovery of new targets and repurposing of drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-99
2. Present to hospital with diagnosis of HF, or

Attending a hospital clinic for management of HF within 6/12 of an episode of decompensated heart failure* which either:

* Resulted in a hospital admission (primary diagnosis) or
* Was treated in out-patient clinic * Appropriate symptoms and signs of HF, confirmed by PI when necessary

Exclusion Criteria:

1. HF primary due to severe valve disease
2. The primary diagnosis is an Acute coronary syndrome (ACS) which has resulted in a transient episode of Acute pulmonary oedema (APO) (Note: Patients with a troponin rise noted during the index admission, but in whom the main presentation is considered clinically to the HF will be included)
3. End stage renal failure (eGFR < 15ml/min/m2) or is receiving or planned to receive renal replacement therapy.
4. Other specific subgroups of HF (Including constrictive pericarditis, complex adult congenital heart disease, hypertrophic cardiomyopathy, eosinophilic myocarditis, cardiac amyloid and acute chemotherapy-induces cardiomyopathy)
5. Isolated right heart failure** (combined right and left heart failure will be included). (Secondary to severe lung disease or pulmonary hypertension)
6. Life threatening co-morbidity with a life expectancy of < 1 year
7. Inability to provide informed consent
8. The patient is unable to comply with study protocol requirements
9. The patient is participating in another clinical research trial(only if that study precludes involvement in an observational study)
10. The patient has declined to participate

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 800 diagnosed heart failure patient will be recruited from primary care clinic, outpatient clinics and hospital ward from Singapore (NUHCS, NHCS, TTSH, CGH, KTPH, SGH).
  800 healthy volunteer control.
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event. | 3 Year

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lam, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No